CLINICAL TRIAL: NCT07399860
Title: Effect of Internal Anal Sphincter Botulinum Toxin A Injection 7 Days Before Hemorrhoidectomy on Postoperative Pain: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Trial
Brief Title: Botulinum Toxin A Before Hemorrhoidectomy to Prevent Postoperative Pain
Acronym: BoTo-HEM
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Lomonosov Moscow State University Medical Research and Educational Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: BoTo-HEM RCT
Record Dates: First submitted 2026-01-20; First posted 2026-02-10 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Hemorrhoids; Postoperative Pain
Keywords: Hemorrhoidectomy; Botulinum toxin; Postoperative pain; Anal sphincter spasm
MeSH Terms: conditions — Hemorrhoids; Pain, Postoperative | interventions — Botulinum Toxins, Type A; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Preoperative Botulinum Toxin A Injection (Experimental): Participants receive a preoperative injection of botulinum toxin type A into the internal anal sphincter seven days prior to excisional hemorrhoidectomy, in addition to standard surgical treatment.
  Interventions: Drug: Botulinum toxin type A
- Preoperative Placebo Injection (Placebo Comparator): Participants receive a preoperative injection of normal saline into the internal anal sphincter seven days prior to excisional hemorrhoidectomy, in addition to standard surgical treatment.
  Interventions: Drug: Saline (0.9% NaCl)

INTERVENTIONS:
Drug: Botulinum toxin type A — Participants receive a single preoperative injection of botulinum toxin type A into the internal anal sphincter. The injection is administered seven days prior to excisional hemorrhoidectomy. Botulinum toxin type A is injected in divided doses at predefined points of the internal anal sphincter using standard technique. The intervention is performed once and no repeat injections are planned.
  Other Names: botox; BTX-A
  Arms: Preoperative Botulinum Toxin A Injection
Drug: Saline (0.9% NaCl) — Participants receive a single preoperative injection of normal saline into the internal anal sphincter. The injection is administered seven days prior to excisional hemorrhoidectomy. Normal saline is injected in divided doses at the same predefined points and using the same technique and injection volume as in the experimental group. The intervention is performed once, with no repeat injections planned.
  Arms: Preoperative Placebo Injection

SUMMARY:
Hemorrhoidectomy is an effective surgical treatment for advanced hemorrhoidal disease but is often associated with significant postoperative pain, which may delay recovery. One of the main contributors to pain after hemorrhoidectomy is spasm and increased tone of the internal anal sphincter.

This randomized, double-blind, placebo-controlled clinical trial evaluates whether preoperative injection of botulinum toxin type A into the internal anal sphincter, performed seven days before hemorrhoidectomy, can reduce postoperative pain compared with placebo. Adult patients with grade III-IV hemorrhoids scheduled for excisional hemorrhoidectomy will be randomized to receive either botulinum toxin A or saline injection prior to surgery.

Postoperative pain intensity, analgesic consumption, complications, functional outcomes, and patient satisfaction will be assessed during the first 30 days after surgery.

DETAILED DESCRIPTION:
This multicenter, randomized, double-blind, placebo-controlled trial is designed to investigate the effect of preoperative botulinum toxin type A injection into the internal anal sphincter on postoperative pain following excisional hemorrhoidectomy.

Eligible adult patients with symptomatic grade III-IV hemorrhoids will be randomized in a 1:1 ratio to receive either botulinum toxin type A or placebo injection seven days prior to surgery. Botulinum toxin A will be injected into the internal anal sphincter in four quadrants using a standardized technique, while the control group will receive an identical volume of normal saline. Both patients and surgeons performing hemorrhoidectomy, as well as outcome assessors, will be blinded to treatment allocation.

All participants will subsequently undergo open or closed hemorrhoidectomy using standardized surgical and perioperative care protocols. Postoperative pain will be assessed using a visual analogue scale during the first seven postoperative days. Secondary outcomes include analgesic consumption, postoperative complications, length of hospital stay, transient fecal incontinence, time to first bowel movement, readmissions, and patient-reported satisfaction within 30 days after surgery.

The study aims to determine whether preoperative chemical sphincter relaxation with botulinum toxin A can improve postoperative recovery and reduce pain following hemorrhoidectomy.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years, male and female
* Symptomatic grade III-IV hemorrhoidal disease (Goligher), refractory to conservative treatment
* Scheduled for open (Milligan-Morgan) or closed (Ferguson) hemorrhoidectomy

Exclusion Criteria:

* Known hypersensitivity to botulinum toxin A, human albumin, or local anesthetics.
* Neuromuscular junction disorders (e.g., myasthenia gravis, Lambert-Eaton syndrome).
* Use of aminoglycosides or other agents interfering with neuromuscular transmission within 14 days.
* Coagulopathy or ongoing anticoagulant therapy not suitable for perioperative interruption.
* Active anorectal infection, fissure, abscess, or inflammatory bowel disease in the active phase.
* Previous anal sphincter surgery or baseline fecal incontinence.
* Pregnancy or breastfeeding.
* ASA ≥ III or significant systemic disease compromising anesthesia or wound healing.
* Participation in another interventional clinical trial within 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 292 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative Pain Intensity Within the First 7 Days After Hemorrhoidectomy | Postoperative days 1-7
  Postoperative pain intensity assessed using a 100-mm visual analogue scale (VAS). Daily pain scores are recorded and used to calculate the area under the curve (AUC) over postoperative days 1-7 for comparison between study groups.

SECONDARY OUTCOMES:
Total opioid consumption within 72 hours postoperatively | Within 72 hours after surgery (postoperative hours 0-72)
  Total postoperative opioid consumption expressed in morphine equivalents (mg) measured within the first 72 hours after surgery. Opioid use is recorded and compared between the botulinum toxin type A group and the placebo group.
Length of hospital stay | From day of surgery until hospital discharge (up to 30 days postoperatively)
  Length of postoperative hospital stay measured in days, calculated from the day of surgery to the day of hospital discharge, and compared between the botulinum toxin type A group and the placebo group.
Incidence of postoperative complications within 30 days | Within 30 days after surgery
  Incidence of postoperative complications occurring within 30 days after surgery, classified according to the Clavien-Dindo classification, and compared between the botulinum toxin type A group and the placebo group.
Transient fecal incontinence rates assessed by Wexner score | Postoperative days 14 and 30
  Transient fecal incontinence assessed using the Wexner score to evaluate severity and frequency of symptoms, and compared between the botulinum toxin type A group and the placebo group.
Readmission or unplanned medical visits within 30 days | Within 30 days postoperatively
  Hospital readmission or unplanned medical visits occurring within 30 days after surgery, compared between the botulinum toxin type A group and the placebo group.
Pain during defecation assessed by VAS | Postoperative days 1, 3, and 7
  Pain intensity during defecation assessed using the Visual Analog Scale (VAS) and compared between the botulinum toxin type A group and the placebo group.
Time to first bowel movement | From day of surgery until first bowel movement (up to hospital discharge, maximum 7 days)
  Time to first bowel movement measured in hours and compared between the botulinum toxin type A group and the placebo group.
Patient satisfaction score | Postoperative day 30
  Patient satisfaction assessed using a numeric rating scale from 0 to 10, where higher scores indicate greater satisfaction. Scores are compared between the botulinum toxin type A group and the placebo group.

CONTACTS AND LOCATIONS:
Overall Officials: Tatiana Garmanova, MD, PhD, Study Director — Lomonosov Moscow State University Medical Research and Educational Center

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to institutional and ethical restrictions and because no data-sharing plan is specified in the study protocol.

REFERENCES:
- [Result] Lie H, Lukito PP, Sudirman T, Purnama AA, Sutedja R, Setiawan A, Jeo WS, Irawan A, Satriya W, Koerniawan HS, Hariyanto TI. Utility of botulinum toxin injection for post-operative pain management after conventional hemorrhoidectomy: a systematic review and meta-analysis of clinical trials. Scand J Gastroenterol. 2023 Feb;58(2):116-122. doi: 10.1080/00365521.2022.2116292. Epub 2022 Sep 1. PMID 36048469
- [Result] Patti R, Arcara M, Bonventre S, Sammartano S, Sparacello M, Vitello G, Di Vita G. Randomized clinical trial of botulinum toxin injection for pain relief in patients with thrombosed external haemorrhoids. Br J Surg. 2008 Nov;95(11):1339-43. doi: 10.1002/bjs.6236. PMID 18844269
- [Result] Jin, J., Unasa, H., Bahl, P. et al. Can Targeting Sphincter Spasm Reduce Post-Haemorrhoidectomy Pain? A Systematic Review and Meta-Analysis. World J Surg 47, 520-533 (2023). https://doi.org/10.1007/s00268-022-06807-3
- [Result] Quinn R, Jamsari G, Albayati S. Botulinum toxin injection for management of post-haemorrhoidectomy pain: an updated systematic review and meta-analysis of randomised clinical trials. Tech Coloproctol. 2025 Apr 7;29(1):96. doi: 10.1007/s10151-025-03137-z. PMID 40192825
- [Result] Sirikurnpiboon S, Jivapaisarnpong P. Botulinum Toxin Injection for Analgesic Effect after Hemorrhoidectomy: A Randomized Control Trial. J Anus Rectum Colon. 2020 Oct 29;4(4):186-192. doi: 10.23922/jarc.2020-027. eCollection 2020. PMID 33134600
- [Result] Yaghoobi Notash A, Sadeghian E, Heshmati A, Sorush A. Effectiveness of Local Botulinum Toxin Injection for Perianal Pain after Hemorrhoidectomy. Middle East J Dig Dis. 2022 Jul;14(3):330-334. doi: 10.34172/mejdd.2022.291. Epub 2022 Jul 30. PMID 36619264
- [Result] Patti R, Almasio PL, Muggeo VM, Buscemi S, Arcara M, Matranga S, Di Vita G. Improvement of wound healing after hemorrhoidectomy: a double-blind, randomized study of botulinum toxin injection. Dis Colon Rectum. 2005 Dec;48(12):2173-9. doi: 10.1007/s10350-005-0179-5. PMID 16400513
- [Result] Davies J, Duffy D, Boyt N, Aghahoseini A, Alexander D, Leveson S. Botulinum toxin (botox) reduces pain after hemorrhoidectomy: results of a double-blind, randomized study. Dis Colon Rectum. 2003 Aug;46(8):1097-102. doi: 10.1007/s10350-004-7286-6. PMID 12907905